CLINICAL TRIAL: NCT05313256
Title: Alkalinization of Adrenalized Lidocaine in Extending Epidural Analgesia for Extremely Urgent Cesarean Section During Labor: a Randomized Controlled Trial.
Brief Title: Quick Epidural Top-up with Alkalinized Lidocaine for Emergent Caesarean Delivery
Acronym: QETAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2021/36
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Obstetric Labor Complications
Keywords: epidural analgesia; caesarean section; sodium bicarbonate; local anesthetics; obstetric labor; alkalinization; extremely urgent
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): In this arm patients will receive for epidural extension a Lidocaine epinephrine buffered with sodium bicarbonate.
  Interventions: Drug: Lidocaine epinephrine buffered with sodium bicarbonate
- Comparator group (Active Comparator): In this arm patients will receive for epidural extension only Lidocaine epinephrine.
  Interventions: Drug: Lidocaine epinephrine

INTERVENTIONS:
Drug: Lidocaine epinephrine buffered with sodium bicarbonate — When an extremely urgent fetal extraction by caesarean section is decided, the patient will be randomized. An epidural top-up will then be performed with Lidocaine epinephrine buffered with sodium bicarbonate.
  Arms: Experimental group
Drug: Lidocaine epinephrine — When an extremely urgent fetal extraction by caesarean section is decided, the patient will be randomized. An epidural top-up will then be performed with Lidocaine epinephrine.
  Arms: Comparator group

SUMMARY:
Prospective randomized study comparing the use of lidocaine 2% with epinephrine buffered with sodium bicarbonate and lidocaine 2% with epinephrine as epidural top-up for extremely urgent cesarean section during labour.

DETAILED DESCRIPTION:
General anesthesia in pregnant women remains burdened by a significant maternal-fetal morbidity and mortality. An increased risk of orotracheal intubation difficulty, gastric inhalation syndrome and neonatal respiratory depression is described.

The rate of epidural analgesia during labor is about 85% in France. In addition to the comfort provided, epidural analgesia allows emergency Caesarean sections to be performed by converting epidural analgesia to epidural anesthesia, a technique known as "epidural extension" or "epidural top-up". The effectiveness and the time necessary to obtain this surgical anesthesia depends on the protocols used and determines the possibility of performing fetal extractions, even the most urgent ones, without resorting to general anesthesia.

We define an extremely urgent cesarean delivery as a delivery required in the event of an immediate threat to maternal or fetal vital prognosis, with a target of less than 15 minutes between the extraction decision time and birth.

In France, the latest recommendations date from 2007 and recommend the practice of epidural extension with 15 to 20 ml of 2% adrenaline lidocaine. With this technique, surgical anesthesia is typically obtained within 10 to 15 minutes. This time remains too long in certain obstetrical emergency situations, notably extremely urgent cesarean sections, which require frequent recourse to general anesthesia to compensate for this length of nerve block installation.

The alkalinization of local anesthetics with sodium bicarbonate has been experimentally studied since the 1970s and makes it possible to accelerate the time of action of local anesthetics. Alkalinization of local anesthetics is practiced in 35% of epidural extensions in Denmark and 12% of epidural extensions in the United Kingdom.

Since 2016, this technique has been used in the anesthesia departments of maternity units of Bayonne and Bordeaux hospitals. In the former, a retrospective study of 51 cases from January 2019 to July 2019 showed a decrease of more than 80% in the rate of recourse to general anesthesia in extremely urgent caesarean sections (4/4 vs 0/7) and a 50% decrease in the time required to obtain adequate epidural anesthesia (5 min vs 10 min).

The main objective of the current prospective study is to prospectively confirm the decrease in the use of general anesthesia in extremely urgent cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, affiliated to social security
* Informed consent signed by the participant and the investigating physician at the latest after the therapeutic intervention
* Initial indication for vaginal delivery
* Benefiting from emergency caesarean section during labour for fetal extraction with a maximum 15-minute decision-to-delivery delay (i.e. extremely urgent caesarean section)

Exclusion Criteria:

* Opposition to participation in research before delivery
* Refusal or impossibility of informed consent
* Lack of understanding or significant language barrier
* Initial indication for general anaesthesia defined by the following situations: non-functional epidural analgesia, altered consciousness, eclampsia, suspicion of amniotic embolism, confirmed or suspected severe haemorrhage occurring before birth
* Contraindication to the use of the products defined in the protocol : adrenalized lidocaine ; sodium bicarbonate.
* Persons placed under judicial protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Resort to general anaesthesia | 15 minutes after inclusion
  Resort to general anaesthesia for insufficient analgesia after epidural extension for extremely urgent caesarean section.

SECONDARY OUTCOMES:
Delay between fetal extraction decision and birth | Between inclusion and birth
  Minutes between the decision to extract the fetus by the obstetrical team and the clamping of the umbilical cord
Delay between fetal extraction decision and incision | Between inclusion and cesarean section
  Minutes between the decision to extract the fetus by the obstetrical team and the surgical incision
Maternal complications | up to 24 hours after inclusion
  Maternal complications after epidural top-up, including nausea-vomiting in the peroperative and postoperative period, desaturation episode, difficult orotracheal intubation, bronchial inhalation syndrome, hypotensive episode before fetal extraction, extended sensory or motor block.
Complementary medicines | Between inclusion and cesarean section
  Use and characterization of complementary medicines necessary for maternal well-being during caesarean section.
Postpartum hemorrhage | up to 24 hours after inclusion
  Postpartum hemorrhage (blood loss of more than 500 ml)
Paediatric wellness | at birth
  Paediatric wellness criteria (umbilical cord pH less than 7.0 ; umbilical cord lactate)
Anesthesia level | one hour after surgical incision
  Anesthesia level one hour after surgical incision
Maternal satisfaction | up to 4 hours after inclusion
  Maternal satisfaction regarding analgesia and anesthesia during caesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas LECHAT, Dr, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, Dr, Study Chair — University Hospital, Bordeaux; Karine NOUETTE-GAULAIN, Pr, Study Director — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CH de la Côte Basque, Bayonne
  - CHU de Bordeaux, Bordeaux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lechat T, d'Aprigny T, Henriot J, Arthur J, Sylla D, Benard A, Nouette-Gaulain K. Quick Epidural Top-up with Alkalinized Lidocaine for emergent caesarean delivery (QETAL study): protocol for a randomized, controlled, bicentric trial. Trials. 2023 May 19;24(1):341. doi: 10.1186/s13063-023-07366-1. PMID 37208675